CLINICAL TRIAL: NCT06394297
Title: A Phase I/II Study for Image Guided Stereotactic Body Radiation Therapy Boost for Definitive Treatment of Locally Advanced Cervical Cancer (LACC)
Brief Title: VIBE - Virtual Image Guided Brachytherapy Emulation for Locally Advanced Cervical Cancer (LACC)
Acronym: VIBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Inês Antunes, Principal Investigator, Fundacao Champalimaud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIBE
Record Dates: First submitted 2024-01-10; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; Stereotactic body radiotherapy (SBRT); Stereotactic ablative body radiotherapy (SABR); Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this study must have received or planned to receive 45 to 50 Gray in 25 fractions to pelvis with a simultaneous integrated boost (SIB) of 55 Gray in 25 fractions to metabolic active primary lesion and of 55 Gray in 25 fractions to 62.5 Gray in 25 fractions suspicious nodes of prior external beam radiation therapy. Following completion, patients will receive a boost of 28 Gray in 4 fractions using Image Guided Stereotactic Body Radiation Therapy techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT for cervical cancer (Experimental): SBRT to LACC following whole pelvis external beam radiotherapy
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT to reproduce HDR BT dose distribution in non-operated patients LACC
  Other Names: SABR

SUMMARY:
This study will evaluate the role of SBRT with the aim to reproduce high dose rate brachytherapy (HDR BT) dose distribution by means of external beam radiotherapy in the radical treatment in patients with LACC. The study will employ devices to accurately reproduce pelvic anatomy and mitigate target motion and will make use of real-time online tracking.

DETAILED DESCRIPTION:
This is a phase I/II feasibility study of hypofractionated, image-guided Volumetric Modulated Arc Therapy (VMAT) Stereotactic Body Radiotherapy (SBRT) to LACC with the aim to reproduce HDR BT dose distribution by means of external beam radiotherapy in the radical treatment in patients with LACC. The study will employ devices to accurately reproduce pelvic anatomy and mitigate target motion and will make use of real-time online tracking.

Eligible patients who consent to participate in the current study will receive 4 image-guided SBRT sessions to a prescription of 7 Gray per fraction to the LACC (HR-CTV) following whole pelvis external beam radiotherapy.

SBRT will start within one week after whole pelvis external beam radiotherapy. The study will enroll a total of 30 patients. After treatment, patients will be followed-up at 1 month, at 3 months (+/- 1 week), at 6 months (+/- 4 weeks), and then every 6 months (+/- 6 weeks) until the end of the 3rd year, then annually until the 5th year.

The equivalence of outcome and toxicity will be measured by comparing the data obtained in the study to literature data regarding the standard modality of brachytherapy. Patients' oncological outcomes, toxicity and quality of life data will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the uterine cervix suitable for curative treatment with definitive radio-chemotherapy
* Biopsy proven showing squamous-cell carcinoma, adenocarcinoma or adeno-squamous cell carcinoma of the uterine cervix.
* Pelvic MRI.
* MRI and Positron emission tomography (PET-CT) of the retroperitoneal space and abdomen at diagnosis is performed.
* Stage IIB to IVA according to International Federation of Gynecological and Obstetrics (FIGO) and TNM guidelines.
* Planning MRI with the applicator in place for the SBRT boost.
* Para-aortic metastatic nodes below L1-L2 are allowed.
* Study specific signed patient informed consent.

Exclusion Criteria:

* Other primary malignancies except carcinoma in situ of the cervix and basal cell carcinoma of the skin.
* Small cell neuroendocrine cancer, melanoma and other rare cancers in the cervix.
* Metastatic disease above and beyond the retroperitoneal paraaortic L1-L2 interspace.
* Previous pelvic or abdominal radiotherapy.
* Previous total or partial hysterectomy.
* Contra-indications to MRI.
* Severe psychiatric condition.
* Severe, active co-morbidity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Dosimetric Feasibility of SBRT boost | through study completion, an average of 3 year
  Fulfillment of protocol dosimetrical endpoints and constraints
reproducibility of SBRT boost | Accuracy of treatment delivery will be measured during the 15 minutes of treatment delivery time
  anatomical accuracy will be confirmed with image guided (CBCT) and online tracking will guarantee a limit of 2mm threshold
Inter/intra fractional target motion | during the 15 minutes of treatment delivery time
  3D deviations recorded in CBCT images and electromagnetic recording
Adverse Events | through study completion, an average of 3 years
  Treatment related side effects based on CTCAE V5.0
Local control | through study completion, an average of 3 years
  Free from loco-regional relapse

SECONDARY OUTCOMES:
Quality of life metrics | through study completion, an average of 3 years
  Change from baseline in European Organisation for Research and Treatment of Cancer quality of life questionnaire C30
Quality of life metrics | through study completion, an average of 3 years
  Change from baseline in European Organisation for Research and Treatment of Cancer quality of life questionnaire N24
Distant Relapse | through study completion, an average of 3 years
  Free from distant relapse

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Greco, MD, Study Director — Fundaçao Champalimaud
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No